CLINICAL TRIAL: NCT01205542
Title: Work Place Adjusted Intelligent Physical Exercise Reducing Musculoskeletal Pain in Shoulder and Neck (VIMS) - Shoulder Function
Acronym: VIMS03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Otto M Poulsen, National Research Centre for the Working Environment
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: VIMS03
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Rehabilitation; Neck Pain; Shoulder Pain; Scapular Dyskinesis; Muscle Activation
MeSH Terms: conditions — Neck Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Training (Experimental): Training of scapular function with strengthening exercises using bodyweight and elastic resistance
  Interventions: Behavioral: Training
- Reference (Active Comparator): Health check and advice to continue ordinary physical activity
  Interventions: Behavioral: Reference

INTERVENTIONS:
Behavioral: Training — Training of scapular function with strengthening exercises using bodyweight and elastic resistance
  Arms: Training
Behavioral: Reference — Health check and advice to continue ordinary physical activity
  Arms: Reference

SUMMARY:
Basic strength training for the neck/shoulder muscles can decrease intensity of neck/shoulder pain, but it is uncertain whether training should focus directly on the upper trapezius - which is most often tender - or on the lower compartments and serratus anterior.

We hypothesize that strengthening exercise for the lower and middle trapezius as well as the serratus anterior will decrease intensity of neck/shoulder pain among office workers

ELIGIBILITY:
Inclusion Criteria:

* employees
* more than 30 days with pain previous year
* pain intensity of at least 3 on a scale of 0-10

Exclusion Criteria:

* trauma
* life threatening disease
* pregnanacy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Neck/shoulder pain | December 2010
  Neck/shoulder pain will be assessed by:
  1. self-report (pain intensity)
  2. clinical examination of muscle tenderness

SECONDARY OUTCOMES:
Muscle function | December 2010
  Muscle strength and electromyography assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Roskilde University Center, Roskilde, Denmark

REFERENCES:
- [Derived] Andersen CH, Andersen LL, Mortensen OS, Zebis MK, Sjogaard G. Protocol for shoulder function training reducing musculoskeletal pain in shoulder and neck: a randomized controlled trial. BMC Musculoskelet Disord. 2011 Jan 14;12:14. doi: 10.1186/1471-2474-12-14. PMID 21235752
- See also: Related Info — http://www.arbejdsmiljoforskning.dk